CLINICAL TRIAL: NCT03063255
Title: Comparison of Obturator Nerve Blockade and Neuromuscular Blockade for the Prevention of Adductor Spasm in Patients Undergoing Transurethral Resection of Bladder Tumors.
Brief Title: Comparison of Obturator Nerve Blockade and Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201601962 -V; OCR18950 (Other: University of Florida)
Record Dates: First submitted 2017-02-08; First posted 2017-02-24 (Actual); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Cancer of Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mepivacaine; Neuromuscular Blockade; Rocuronium

STUDY DESIGN:
Intervention Model Description: Sixty subjects with be randomized to the obturator block or neuromuscular block arm upon enrollment, using randomized permutated blocks of six.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obturator block (Active Comparator): Comparing the incidence of adductor spasm in patients undergoing general anesthesia with obturator block.
  Interventions: Drug: Obturator block
- Neuromuscular block (Active Comparator): Comparing the incidence of adductor spasm in patients undergoing general anesthesia with neuromuscular blocking agents.
  Interventions: Drug: Neuromuscular block

INTERVENTIONS:
Drug: Obturator block — Subjects allocated to the obturator block group will be monitored for the incidence of block and procedure-related adverse events. In addition to clinical observation, a Nerve Integrity Monitor (Medtronic) will be used to detect adductor spasm using continuous electromyography. Electrodes will be placed on the thigh to objectively detect and record instances of adductor spasm. One hour after arrival to post-anaesthesia care unit (PACU) or when discharge criteria are met (whichever comes first), repeat dynamometer measurements and TUG tests will be performed. Patients will be called 24-48 hours post procedure to inquire about falls or evidence of nerve injury, as well as patient satisfaction.
  Other Names: Ultrasound guided nerve block anesthetic; Mepivacaine; Pajunk SonoPlex needle
  Arms: Obturator block
Drug: Neuromuscular block — Subjects allocated to the neuromuscular block group will be monitored for the incidence of block and procedure-related adverse events. In addition to clinical observation, a Nerve Integrity Monitor (Medtronic) will be used to detect adductor spasm using continuous electromyography. Electrodes will be placed on the thigh to objectively detect and record instances of adductor spasm. One hour after arrival to PACU or when discharge criteria are met (whichever comes first), repeat dynamometer measurements and TUG tests will be performed. Patients will be called 24-48 hours post procedure to inquire about falls or evidence of nerve injury, as well as patient satisfaction.
  Other Names: Paralysis of the affected skeletal muscles anesthetic; Rocuronium
  Arms: Neuromuscular block

SUMMARY:
Patients diagnosed with posterolateral bladder tumors will be invited to participate in the study. Subjects will be randomized to receive an ultrasound-guided obturator block or a neuromuscular blocking agent after the induction of general anesthesia in an attempt to block the obturator reflex during surgery.

DETAILED DESCRIPTION:
The purpose of this research is to compare the incidence of adductor spasm in patients undergoing general anesthesia with neuromuscular blocking agents versus obturator block. Transurethral resection of bladder tumor(s) (TURBT) is a commonly performed procedure to diagnose and treat bladder cancer. The obturator nerve is located lateral to the bladder wall in the pelvis prior to innervating the adductor muscles of the thigh. Depending on the location of the tumor(s), electrocautery or surgical stimulation may result in stimulation of the obturator nerve, resulting in adduction of the leg, which is called the adductor reflex or spasm. This may occur violently and unexpectedly, and result in bladder perforation, bleeding, or cancer dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Planned TURBT for unilateral or bilateral posterolateral bladder tumors
* Ability to understand and provide informed consent

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* True allergy, not sensitivity, to local anesthetics
* True allergy, not sensitivity, Propofol
* True allergy, not sensitivity, general anesthetic agents
* Pregnancy
* Severe hepatic impairment
* Evidence of infection at or near the proposed needle insertion site
* Any sensorimotor deficit of the lower extremity, whether acute or chronic
* Inability to walk without assistance
* Lower extremity joint replacement surgery in the preceding six months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José R Soberón, MD, Principal Investigator — Malcom Randall VA Medical Center; Benjamin Canales, MD, Principal Investigator — University of Florida
Locations (1):
- Malcom Randall VA Medical Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soberon JR, Awoniyi CA, Perez MA, Vasilopoulos T, Canales BK. Obturator Nerve Blockade vs. Neuromuscular Blockade for the Prevention of Adductor Spasm in Patients Undergoing Transurethral Resection of Bladder Tumors: A Randomized Controlled Trial. Pain Med. 2021 Jun 4;22(6):1253-1260. doi: 10.1093/pm/pnaa448. PMID 33537703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled was on 04/25/2017 and the last subject enrolled was on 6/11/2019. All subjects were enrolled at the Malcom Randall VAMC.
Period: Overall Study
Arm/Group | Obturator Block | Neuromuscular Block
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: data entry error, one subject was withdrawn and demographic data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obturator Block | Neuromuscular Block | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.3) | 72.2 (6.3) | 71.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — One subject was withdrawn as a significant adverse event occurred. The patient was enrolled in the study and suffered a cardiac arrest after induction of general anesthesia. The etiology was likely myocardial ischemia from cardiac stent thrombosis (unrelated to the study intervention). Only baseline demographic information was collected for the study on this withdrawn patient.
  participants
    United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Incidence of Intraoperative Adductor Spasm
Description: Nerve Integrity Monitor will be used to detect adductor spasm and below are listed the numbers or patients with increased incidence of adductor spasm.
Time Frame: intraoperative
Population: Data entry error correction, one patient withdrawn and only demographic information collected
Measure: Count of Participants; unit: Participants
Arm/Group | Obturator Block | Neuromuscular Block
Number analyzed (Participants) | 29 | 30
Participants | 1 | 5

2. Secondary Outcome: Number Patients With Increased Risk of Falling
Description: Based on TUG time measurements of patients below are the numbers of patients with an increased risk of falling.
Time Frame: Changes from baseline (pre-op) to 72 hours post-operative
Population: Data entry error correction, one patient withdrawn and only demographic information collected
Measure: Number; unit: participants
Arm/Group | Obturator Block | Neuromuscular Block
Number analyzed (Participants) | 29 | 30
participants | 28 | 29

3. Secondary Outcome: Number of Patients With Incidence of Leg Weakness
Description: Test the strength of subject's lower extremity muscles on the timed up and go (TUG) test and determine how many patients had increased leg weakness.
Time Frame: Changes from baseline (pre-op) to 72 hours post-operative
Population: Data entry error correction, one patient withdrawn and only demographic information collected
Measure: Count of Participants; unit: Participants
Arm/Group | Obturator Block | Neuromuscular Block
Number analyzed (Participants) | 29 | 30
Participants | 27 | 22

ADVERSE EVENTS:
Time Frame: For the overall study adverse events were recorded over 1 year and 2 months. Each subject was followed for AE's per protocol.
Arm/Group | Obturator Block | Neuromuscular Block
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03063255/Prot_SAP_002.pdf
  • Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03063255/ICF_004.pdf